CLINICAL TRIAL: NCT06257589
Title: A Grounded Theory of Phrenic Nerve Reconstruction for the Treatment of Diaphragm Paralysis - A Biopsychosocial Approach to Surgical Evaluation and Outcomes
Brief Title: A Chart Review to Evaluate the Safety and Efficacy of Phrenic Nerve Reconstruction for the Treatment of Diaphragmatic Paralysis
Status: Active, not recruiting | Type: Observational
Sponsor: Advanced Reconstructive Surgery Alliance (Other Government)
Responsible Party: Principal Investigator, Matthew Kaufman, MD, Head of Phrenic Nerve Reconstructive Surgery., Advanced Reconstructive Surgery Alliance
Other Study IDs: GT-Phase-1
Record Dates: First submitted 2024-01-17; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Diaphragm Issues; Diaphragm; Paralysis, Due to Accidental Section of Phrenic Nerve During Procedure; Breath Shortness; Diaphragmatic Paralysis
Keywords: Grounded Theory; Mixed Methods; Chart Review; Diaphragmatic Paralysis
MeSH Terms: conditions — Paralysis; Dyspnea; Respiratory Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intrathoracic Approach: Patients who have undergone the intrathoracic approach of phrenic nerve reconstruction for the treatment of diaphragmatic paralysis.
  NO INTERVENTION.
- Cervical Approach: Patients who have undergone the cervical approach of phrenic nerve reconstruction for the treatment of diaphragmatic paralysis.
  NO INTERVENTION.

SUMMARY:
A retrospective chart review to evaluate the safety and efficacy of phrenic nerve reconstruction for diaphragmatic paralysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent phrenic nerve reconstructive surgery for the treatment of Diaphragmatic Paralysis.

Exclusion Criteria:

* Age 18 and below.

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent phrenic nerve reconstructive surgery for the treatment of Diaphragmatic Paralysis.
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Radiographic Position of Diaphragm. | Up to 12 Months.
  Radiographic Thoracic Imaging.
Pulmonary Function. | Up to 12 Months.
  Pulmonary Function Test (PFT).

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQoL). | Up to 12 Months.
  SF-36 / RAND Survey.
Safety of Phrenic Nerve Reconstruction for Diaphragmatic Paralysis. | Up to 24 Months.
  AEs related to the procedure reported in the medical chart.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kaufman, MD, Principal Investigator — Advanced Reconstructive Surgery Alliance
Locations (2):
- United States (2):
  - Advanced Reconstructive Surgery Alliance, Red Bank, New Jersey
  - Institute for Advanced Reconstruction, Shrewsbury, New Jersey

IPD SHARING:
Plan to Share IPD: No
No Individual participant data (IPD) will not be shared.

REFERENCES:
- [Background] Kaufman MR, Ferro N, Paulin E. Phrenic nerve paralysis and phrenic nerve reconstruction surgery. Handb Clin Neurol. 2022;189:271-292. doi: 10.1016/B978-0-323-91532-8.00003-3. PMID 36031309
- [Background] Kaufman MR, Chang EI, Bauer T, Rossi K, Elkwood AI, Paulin E, Jarrahy R. Phrenic Nerve Reconstruction for Effective Surgical Treatment of Diaphragmatic Paralysis. Ann Plast Surg. 2021 Sep 1;87(3):310-315. doi: 10.1097/SAP.0000000000002896. PMID 34397519
- [Background] Kaufman MR, Bauer T, Onders RP, Brown DP, Chang EI, Rossi K, Elkwood AI, Paulin E, Jarrahy R. Treatment for bilateral diaphragmatic dysfunction using phrenic nerve reconstruction and diaphragm pacemakers. Interact Cardiovasc Thorac Surg. 2021 May 10;32(5):753-760. doi: 10.1093/icvts/ivaa324. PMID 33432336
- [Background] Kaufman MR, Bauer T, Campbell S, Rossi K, Elkwood A, Jarrahy R. Prospective analysis of a surgical algorithm to achieve ventilator weaning in cervical tetraplegia. J Spinal Cord Med. 2022 Jul;45(4):531-535. doi: 10.1080/10790268.2020.1829417. Epub 2020 Oct 15. PMID 33054689
- [Background] Kaufman MR, Willekes LJ, Elkwood AI, Rose MI, Patel TR, Ashinoff RL, Colicchio AR. Diaphragm paralysis caused by transverse cervical artery compression of the phrenic nerve: the Red Cross syndrome. Clin Neurol Neurosurg. 2012 Jun;114(5):502-5. doi: 10.1016/j.clineuro.2012.01.048. Epub 2012 Feb 24. PMID 22366245
- [Background] Kaufman MR, Elkwood AI, Brown D, Cece J, Martins C, Bauer T, Weissler J, Rezzadeh K, Jarrahy R. Long-Term Follow-Up after Phrenic Nerve Reconstruction for Diaphragmatic Paralysis: A Review of 180 Patients. J Reconstr Microsurg. 2017 Jan;33(1):63-69. doi: 10.1055/s-0036-1588018. Epub 2016 Sep 25. PMID 27665114
- [Background] Kaufman MR, Elkwood AI, Colicchio AR, CeCe J, Jarrahy R, Willekes LJ, Rose MI, Brown D. Functional restoration of diaphragmatic paralysis: an evaluation of phrenic nerve reconstruction. Ann Thorac Surg. 2014 Jan;97(1):260-6. doi: 10.1016/j.athoracsur.2013.09.052. Epub 2013 Nov 19. PMID 24266954
- [Background] Kaufman MR, Elkwood AI, Rose MI, Patel T, Ashinoff R, Saad A, Caccavale R, Bocage JP, Cole J, Soriano A, Fein E. Reinnervation of the paralyzed diaphragm: application of nerve surgery techniques following unilateral phrenic nerve injury. Chest. 2011 Jul;140(1):191-197. doi: 10.1378/chest.10-2765. Epub 2011 Feb 24. PMID 21349932
- [Background] Kaufman MR, Elkwood AI, Rose MI, Patel T, Ashinoff R, Fields R, Brown D. Surgical treatment of permanent diaphragm paralysis after interscalene nerve block for shoulder surgery. Anesthesiology. 2013 Aug;119(2):484-7. doi: 10.1097/ALN.0b013e31829c2f22. No abstract available. PMID 23838708
- [Background] Kaufman MR, Elkwood AI, Aboharb F, Cece J, Brown D, Rezzadeh K, Jarrahy R. Diaphragmatic reinnervation in ventilator-dependent patients with cervical spinal cord injury and concomitant phrenic nerve lesions using simultaneous nerve transfers and implantable neurostimulators. J Reconstr Microsurg. 2015 Jun;31(5):391-5. doi: 10.1055/s-0035-1549159. Epub 2015 Apr 13. PMID 25868155